CLINICAL TRIAL: NCT06549218
Title: Shortening the Path to Rare Disease Diagnosis by Using Newborn Genetic Screening and Digital Technologies (SCREEN4CARE): Genetic Newborn Screening for Rare Diseases Within the Screen4Care Project
Brief Title: Genetic Newborn Screening for Rare Diseases Within the Screen4Care Project
Acronym: SCREEN4CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Innovative Medicines Initiative (Other); Università degli Studi di Ferrara (Other); Ospedale Pediatrico Bambin Gesù (Other); University of Siena (Other); Centre Hospitalier Universitaire Dijon (Other); Real Genix (Unknown); University Hospital Goettingen (Other); Centro Nacional de Análisis Genómico (Unknown); Genoox (Unknown); Schwarzwald-Baar Clinic (Unknown); Municipal Hospital Karlsruhe (Unknown)
Responsible Party: Principal Investigator, Jan Kirschner, Prof. Dr., University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 101034427; NCT06528548 (obsolete NCT alias)
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Newborn Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- newborn screening (Other): All newborns participating in the study will receive a genetic newborn screening for predefined treatable diseases. Newborns participating in the TREAT-panel developing symptoms suggestive of a genetic disease during the first 2 years of life can receive whole genome sequencing.
  Interventions: Diagnostic Test: newborn genetic screening and whole genome sequencing

INTERVENTIONS:
Diagnostic Test: newborn genetic screening and whole genome sequencing — newborn genetic screening (panel of treatable diseases); whole genome sequencing (if newborn develops symptoms suggestive of a genetic disease)

SUMMARY:
The main objective of the genetic newborn screening part of the Screen4Care-project is to shorten the path to rare disease diagnosis and to facilitate early intervention. Therefore, genetic newborn screening for currently treatable rare diseases (TREAT-panel approach) will be offered to families expecting a baby. Whole genome sequencing (WGS) will be offered as additional diagnostic approach to newborns participating in Screen4Care TREAT-panel approach, if they develop symptoms suggestive of a genetic disease.

To evaluate to what extend genetic newborn screening has an impact on participating infants and their families, a follow-up with standardised questionnaires will be performed for all participating families.

ELIGIBILITY:
Inclusion Criteria:

* TREAT-panel:

  * newborns
  * Infants born in one of the participating hospitals and birth centres
  * Informed consent signed by both parents/legal guardian to participate in genetic newborn screening (TREAT-panel)
* Whole genome sequencing:

  * Participation in the TREAT-panel study
  * Symptoms suggestive of a genetic disease within the first 2 years of life
  * Informed consent signed by both parents/legal guardian to participate in genetic newborn screening (TREAT-panel) and the whole genome sequencing

Exclusion Criteria:

* Missing informed consent of parents/legal guardian

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
TREAT-panel | 1 year
  • Percentage of eligible couples who will accept to participate to the genetic newborn screening
TREAT-panel | 1 year
  • Percentage of infants in whom pathogenic or likely pathogenic variants that predict one of the target diseases will be identified
Whole Genome Sequencing | 2 years
  • Percentage of symptomatic patients whom parents will accept to be enrolled in whole genome sequencing
Whole Genome Sequencing | 2 years
  • Percentage of known disease genes where pathogenic variations will be identified by whole genome sequencing in enrolled patients
Whole Genome Sequencing | 2 years
  • Percentage of infants where genetic diagnosis is achieved by whole genome sequencing

SECONDARY OUTCOMES:
TREAT-panel | 1 year
  • Clinical follow-up of infants with positive findings in gNBS
TREAT-panel | 1 year
  • Impact of genetic NBS on parents as assessed by standardized questionnaires
TREAT-panel | 1 year
  • Carrier frequency of recessive diseases (both autosomal and X-linked) and percentage of variants of unknown significance identified through gNBS.
TREAT-panel | 1 year
  • Percentage of study participants who develop symptoms of a genetic disease after negative newborn screening and are diagnosed by whole genome sequencing (aggregated data analysis, not reported to participants)
TREAT-panel | 1 year
  • Impact of positive findings in gNBS on the health care and outcome of study participants
Whole Genome Sequencing | 2 years
  • Percentage of novel disease genes (phenotype discovery) where pathogenic variations will be identified by Whole Genome Sequencing in enrolled patients
Whole Genome Sequencing | 2 years
  • Number of VUS identified in known disease genes
Whole Genome Sequencing | 2 years
  • Number of VUS identified in novel disease genes/phenotypes
Whole Genome Sequencing | 2 years
  • Diagnostic yield of Whole Genome Sequencing compared to genetic newborn screening

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferlini, Professor, Principal Investigator — Unit Medical Genetics, Azienda Ospedaliero-Universitaria Sant'Anna
Locations (6):
- Centre de Génétique et Centre de Référence Anomalies du Développement et Syndromes Malformatifs, Hôpital d'Enfants, Dijon, France
- Clinic for Neuropediatrics and Muscular Diseases, Freiburg University Medical Center, Freiburg im Breisgau, Germany
- Italy (4):
  - Ospedale Pediatrivo Bambino Gesu IRCCS, Rome, Lazio
  - Unit Medical Genetics, Azienda Ospedaliero-Universitaria Sant'Anna, Ferrara
  - Azienda Ospedaliero Universitaria di Modena, Neonatology Unit, Modena
  - San Pietro Fatebenefratelli Hospital, Roma

IPD SHARING:
Plan to Share IPD: No